CLINICAL TRIAL: NCT00137904
Title: Study of Sleep Disorders and Fatigue in Patients With Multiple Sclerosis
Brief Title: Sleep Disorders in Patients With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Other Study IDs: RBM0242
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2006-02-09 (Estimated); Status verified 2005-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; fatigue; sleep disorders
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Fatigue is a frequent and disabling symptom in patients with multiple sclerosis (MS). The pathophysiology of this sign is not fully understood. Some data suggest that the fatigue is associated with sleep disorders. The aim of this study is to determine the polysomnographic parameters in MS patients with fatigue in comparison to MS patients without fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple sclerosis
* Expanded Disability Status Scale score < or = 5
* Fatigue (Modified Fatigue Impact Scale > 45), with a disease duration > 3 months

Exclusion Criteria:

* Depression
* Cognitive disorders
* EDSS > 5
* Epilepsia
* Obesity
* Drug inducing sleep disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Stankoff, MD, PhD, Principal Investigator — CIC-Pitié-Salpêtrière
Locations (1):
- Centre d'Investigation Clinique-Hopital Pitié-Salpêtrière, Paris, France